CLINICAL TRIAL: NCT07324837
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study of the Efficacy and Safety of the Recombinant Non-immunogenic Staphylokinase in Patients With Acute Ischemic Stroke Within 4.5-24 Hours of Symptom Onset (FRIDA-CT)
Brief Title: Single Bolus Non-immunogenic Staphylokinase in Patients With Acute Ischemic Stroke Within 4.5-24 Hours of Symptom Onset
Acronym: FRIDA-CT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Supergene, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FRIDA-CT
Record Dates: First submitted 2025-12-23; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Ischemic Stroke, Acute
Keywords: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-immunogenic staphylokinase (Experimental): The non-immunogenic staphylokinase is given as a single intravenous bolus, 10 mg (within 5-10 seconds) immediately upon randomization regardless patient's bodyweight
  Interventions: Drug: non-immunogenic staphylokinase
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: non-immunogenic staphylokinase — The non-immunogenic staphylokinase is given as a single intravenous bolus, 10 mg (within 5-10 seconds) immediately upon randomization regardless patient's bodyweight
  Other Names: Fortelyzin®
  Arms: Non-immunogenic staphylokinase
Drug: Placebo — Placebo is given as a single intravenous bolus (within 5-10 seconds) immediately upon randomization
  Arms: Placebo

SUMMARY:
Multicenter, double-blind, randomized, placebo-controlled phase III clinical trial. At the clinical sites, patients with acute ischemic stroke within 4.5-24 hours of symptom onset will be randomized to receive a single bolus injection of the recombinant non-immunogenic staphylokinase (Fortelyzin®, LLC "SuperGene", Russia) or placebo.

DETAILED DESCRIPTION:
The current guidelines recommended intravenous thrombolysis as the first-line treatment for acute large vessel occlusion of anterior circulation stroke within 4.5 hours of stroke onset. However, a majority of patients arrive in the hospital outside the 4.5-hour time window, who could not receive intravenous thrombolysis.

In 2020, the non-immunogenic staphylokinase was registered in Russia for the acute ischemic stroke treatment within 4,5 h after the onset of symptoms. In the FRIDA randomized clinical trial the non-immunogenic staphylokinase was non-inferior to alteplase for patients with acute ischaemic stroke. Mortality, symptomatic intracranial haemorrhage, and serious adverse events did not differ significantly between groups. Non-immunogenic staphylokinase is easy to administer with a rapid single bolus of 10 mg regardless patients' bodyweight, simplifying clinical use. In 2024, the non-immunogenic staphylokinase has been included in the updated Russian clinical guidelines for the acute ischemic stroke treatment.

A rapid (10 s) single bolus of the non-immunogenic staphylokinase in patients with acute ischemic stroke may provide significant advantages over a one-hour alteplase administration in the more rapid reperfusion in the first 24 hours after thrombolysis and a greater number of good functional outcomes. It can be assumed that the non-immunogenic staphylokinase usage in patients with acute ischemic stroke outside the 4.5-hour therapeutic window will lead to the restoration of collateral blood flow in the penumbra in comparison with standard medical management.

Therefore, FRIDA-CT trial is aimed to investigate the efficacy and safety of the non-immunogenic staphylokinase within the time window of 4.5-24 hours, wake-up stroke or no witness stroke in patients who had an acute ischaemic stroke with salvageable tissue due to large vessel occlusion.

In the multicenter, double-blind, randomized, placebo-controlled phase III clinical trial patients who had an acute ischaemic stroke due to anterior circulation large vessel occlusion (internal carotid artery, middle cerebral artery M1 and M2 segments) within 4.5-24 hours from last known well (including wake-up stroke and no witness stroke) and with salvageable tissue (ischaemic core volume <70 mL, mismatch ratio ≥1.8 and mismatch volume ≥15 mL) based on CT perfusion or MRI perfusion-weighted imaging (PWI) will be included and randomised to the non-immunogenic staphylokinase, 10 mg (single bolus) regardless patient's bodyweight or placebo group. Patients who are intended for direct thrombectomy will be excluded from the trial. Follow-up period will be 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 years and over;
2. Acute ischemic stroke symptom onset between 4.5 to 24 hours prior to enrolment, including wake-up stroke and unwitnessed stroke, onset time refers to "last-seen normal time";
3. Pre-stroke modified Rankin scale (mRS) score≤1;
4. Internal carotid artery, middle cerebral artery M1 or M2 occlusion confirmed by CT/MRI, internal carotid artery, middle cerebral artery M1 or M2 being responsible for signs and symptoms of acute ischemic stroke;
5. Neuroimaging: target mismatch profile on CT or MRI perfusion: ischemic core volume <70 mL, mismatch ratio≥1.8 and mismatch volume≥15 mL;
6. Alberta Stroke Program Early CT score (ASPECTS) > 6;
7. Baseline National Institutes of Health Stroke Scale (NIHSS) 6-25 (inclusive);
8. The patient is not planned or cannot undergo thrombectomy or intravenous thrombolysis in accordance with the current version of the Clinical Guidelines;
9. Written informed consent from patients or their legally authorized representatives.

Exclusion Criteria:

1. Acute ischemic stroke within 4,5 h after symptom onset;
2. Intended to proceed to endovascular treatment;
3. Known hypersensitivity to the non-immunogenic staphylokinase;
4. Convulsive seizures at the onset of the disease, if there is no certainty that the seizure is a clinical manifestation of acute ischemic stroke;
5. Persistent blood pressure elevation (systolic ≥185 mmHg or diastolic ≥110 mmHg), and the inability to reduce systolic blood pressure below 180 mmHg or diastolic blood pressure below 105 mmHg;
6. Blood glucose <2.8 or >22.2 mmol/L (after blood glucose level correction to the specified values, inclusion of the patient in the study is possible);
7. Neuroimaging (CT, MRI) signs of intracranial hemorrhage, brain tumor, arteriovenous malformation, brain abscess, cerebral aneurysm;
8. Subarachnoid hemorrhage;
9. Major bleeding currently or within the past 6 months;
10. Surgery on the brain or spinal cord in the last 2 months;
11. Punctures of non-compressible arteries and veins in the last 7 days;
12. Gastrointestinal or genitourinary bleeding in the last 3 weeks. Confirmed exacerbations of gastric ulcer and duodenal ulcer in the last 3 months;
13. Platelet count below 100,000/mm3;
14. Previous stroke or severe traumatic brain injury within 3 months;
15. Unable to perform CT or MRI;
16. History of hemorrhagic stroke or stroke of unspecified genesis;
17. Multiple arterial occlusion (bilateral MCA occlusion, MCA occlusion accompanied with basilar occlusion);
18. Concomitant use of indirect oral anticoagulants (warfarin) with INR > 1.7;
19. Taking direct anticoagulants (heparin, heparinoids) in the previous 48 hours with an APTT value above normal;
20. Taking new oral anticoagulants in the previous 48 hours with a thrombin time value above normal and the impossibility of administering the specific antagonist idarucizumab (for dabigatran) or the presence of anti-Xa activity (for rivaroxaban, apixaban and edoxaban).
21. Severe liver disease, including liver failure, liver cirrhosis, portal hypertension (with esophageal varices), active hepatitis;
22. Acute pancreatitis;
23. Bacterial endocarditis, pericarditis;
24. Arterial aneurysms, malformations of arteries and veins. Suspected dissecting aortic aneurysm;
25. Cancer with an increased risk of bleeding;
26. Major surgeries or severe injuries within the last 14 days, minor surgeries or invasive procedures within the last 10 days;
27. Prolonged or traumatic cardiopulmonary resuscitation (more than 2 minutes);
28. Hemorrhagic diathesis, including renal and hepatic failure;
29. Data on bleeding or acute trauma (fracture) at the time of examination;
30. Pregnant women, nursing mothers, or reluctant to use effective contraceptive measures during the period of trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Good functional outcome | 90 days
  The number of patients with good functional outcome defined as an mRS score 0-1 at 90 days

SECONDARY OUTCOMES:
Ordinal distribution of mRS | 90 days
  Ordinal distribution of mRS at 90 days
Functional independence outcome | 90 days
  The number of patients with functional independence defined by an mRS score 0-2 point at 90 days
NIHSS change from baseline | 7-14 days
  NIHSS median change from baseline on discharge
The rate of improvement on reperfusion | 24 hours
  The number of patients with recanalization of 2 and 3 points on the arterial occlusion scale (rAOL) 24 hours after drug administration according to CT (MRI) angiography, where 0 points - complete occlusion, 3 points - complete recanalization.
All-cause mortality | 90 days
  Rate of all-cause mortality within 90 days
Poor functional outcome | 90 days
  The number of patients with poor functional outcome defined by an mRS score 5-6 point at 90 days

OTHER OUTCOMES:
Hemorrhagic transformation | 24 hours
  Rate of hemorrhagic transformation according to The Heidelberg Bleeding Classification within 24 hours
Symptomatic intracranial hemorrhage | 24 hours
  Rate of symptomatic intracranial hemorrhage (sICH) (as defined by The European Cooperative Acute Stroke Study III criteria [ECASSIII] and Safe Implementation of Thrombolysis in Stroke-Monitoring Study [SITS-MOST]) within 24 hours
Major bleeding | 90 days
  Rate of major bleeding at 90 days (as defined by the Bleeding Academic Research Consortium (BARC) scale: type 3 and type 5)
Serious adverse events (SAEs) | 90 days
  Rate of serious adverse events (SAEs) within 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Nikolay A. Shamalov, MD, prof, Principal Investigator — Federal Center for Brain and Neurotechnology of the Federal Medical and Biological Agency of Russia; Sergey S. Markin, MD, prof, Study Director — LLC "SuperGene"
Locations (15):
- Russia (15):
  - Ryazan Regional Clinical Hospital, Ryazan, Ryazan Oblast
  - Altai Regional Clinical Hospital, Barnaul
  - Chelyabinsk Regional Clinical Hospital No. 3, Chelyabinsk
  - Irkutsk Regional Clinical Hospital, Irkutsk
  - Kaluga Regional Clinical Hospital, Kaluga
  - Interregional Clinical and Diagnostic Center, Kazan'
  - S.V. Ochapovsky Research Institute - Regional Clinical Hospital No. 1, Krasnodar
  - N.I. Pirogov Russian National Research Medical University, Moscow
  - V.I. Voynov Orenburg Regional Clinical Hospital, Orenburg
  - Leningradskaya Regional Clinical Hospital, Saint Petersburg
  - Sergiev Posad District Hospital, Sergiyev Posad
  - Tver Regional Clinical Hospital, Tver'
  - Ulyanovsk Regional Clinical Hospital, Ulyanovsk
  - City Clinical Hospital of Emergency Medical Care No. 25, Volgograd
  - Sverdlovsk Regional Clinical Hospital No. 1, Yekaterinburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gusev EI, Martynov MY, Nikonov AA, Shamalov NA, Semenov MP, Gerasimets EA, Yarovaya EB, Semenov AM, Archakov AI, Markin SS; FRIDA Study Group. Non-immunogenic recombinant staphylokinase versus alteplase for patients with acute ischaemic stroke 4.5 h after symptom onset in Russia (FRIDA): a randomised, open label, multicentre, parallel-group, non-inferiority trial. Lancet Neurol. 2021 Sep;20(9):721-728. doi: 10.1016/S1474-4422(21)00210-6. PMID 34418399
- [Result] Shamalov NA, Martynov MY, Yarovaya EB, Chefranova ZY, Kutsenko VA, Semenov AM, Ivanov SV, Semenov MP, Markin SS, Gusev EI; FORPI Study Group. Thrombolysis With the Non-Immunogenic Staphylokinase for Acute Ischemic Stroke in the FORPI Registry: An Observational Study. Stroke. 2026 Feb;57(2):394-403. doi: 10.1161/STROKEAHA.125.051115. Epub 2025 Nov 26. PMID 41293810